CLINICAL TRIAL: NCT06357325
Title: Determining The Opinions of Women Living In The Earthquake Zone On The Physical and Psychosocial Problems After The 2023 Kahramanmaraş Earthquake
Brief Title: 2023 Problems Faced by Women Earthquake Survivors in Kahramanmaraş
Status: Completed | Type: Observational
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Özen İnam, Asst.Prof.Dr, Maltepe University
Other Study IDs: E-74555795-050.01.04-52290
Record Dates: First submitted 2024-03-21; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Psychosocial Problem; Nurse-Patient Relations; Disaster; Personality; Gender
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: The study was designed as a qualitative (semi-structured) study. The population of the study consisted of women affected by the 2023 Kahramanmaraş-Pazarcık fault line centred earthquake. The sample consisted of women aged 18 years and older who lived in Hatay, Kahramanmaraş and Adana provinces during and after the earthquake and who agreed to participate in the study.
  Data collection method: Participants were recruited using snowball sampling. The study plan was given to the people living in the earthquake zone who were reached by the researcher. Then the participants were reached by informing each other about the study. Interviews with the participants were conducted by telephone interviews to avoid spatial, temporal and transport constraints. The study "themes" were formed according to the responses to the pre-structured open-ended questions.
  Interventions: Other: a qualitative study.

INTERVENTIONS:
Other: a qualitative study. — Before the interview process began, an interview form was created in accordance with the study design. In the study, care was taken to use open-ended general questions that would allow the participant to provide detailed information on the subject and did not require short answers such as short and clear questions, multiple choice questions, and yes-no questions.
  For the analysis and reporting phase, an introduction was made in the form of a conversation with the participant before starting the interview, and then the interview was started if the participant was available. During the transcription phase, the questions were asked during the interview in such a way as to allow the participant to express themselves in detail without any direction or comment. The interview was conducted individually by calling each woman by telephone. During the interview, the researcher transcribed the interviewee's sentences exactly as she expressed them.

SUMMARY:
Objective:

This study was conducted to evaluate the opinions of earthquake victims about the problems affecting women's health physically and psychosocially after the 2023 Kahramanmaraş earthquake.

Method:

The study was designed in a qualitative type (semi-structured). The population of the study consisted of women affected by the 2023 Kahramanmaraş-Pazarcık earthquake. 15 women were interviewed.

DETAILED DESCRIPTION:
Study Design The study was designed as a qualitative (semi-structured) study. The population of the study consisted of women affected by the 2023 Kahramanmaraş-Pazarcık fault line centred earthquake. The sample consisted of women aged 18 years and older who lived in Hatay, Kahramanmaraş and Adana provinces during and after the earthquake and who agreed to participate in the study.

Inclusion Criteria Being over 18 years of age, being mentally healthy, speaking Turkish, being in the earthquake zone during the earthquake.

Data collection method: Participants were recruited using snowball sampling. The study plan was given to the people living in the earthquake zone who were reached by the researcher. Then the participants were reached by informing each other about the study. Interviews with the participants were conducted by telephone interviews to avoid spatial, temporal and transport constraints. The study "themes" were formed according to the responses to the pre-structured open-ended questions.

Study questions:

* What are the demographic changes experienced by women after the earthquake?
* What are the physical problems experienced by women after the earthquake?
* What are the psychological/spiritual problems experienced by women after the earthquake?
* What are the needs and difficulties of women after the earthquake?
* What are the difficulties experienced by women in social life after the earthquake? Data collection tools: A semi-structured interview form, developed by the researcher through literature review, was used as a data collection tool. The form consists of 3 sections: personal information, changes experienced during the earthquake and problems of being a woman during the earthquake.

The first part of the form consists of personal information (age, occupation, marital status, number of children, spouse's occupation, educational status, income status).

The second part consists of questions about changes experienced after the earthquake (loss of first-degree relatives, change in income status, living in a house/tent/container).

The third part consists of open-ended questions on opinions about life after the earthquake (changes in life in general; moving, changing jobs, etc.; problems of being a woman; hygiene, etc.).

The interview form consists of 18 questions, the last 5 of which are open questions.

The interview was conducted individually with each woman and each interview lasted approximately 40 minutes.

Data Analysis Before the interview process began, an interview form was created in accordance with the study design. In the study, care was taken to use open-ended general questions that would allow the participant to provide detailed information on the subject and did not require short answers such as short and clear questions, multiple choice questions, and yes-no questions.

For the analysis and reporting phase, an introduction was made in the form of a conversation with the participant before starting the interview, and then the interview was started if the participant was available. During the transcription phase, the questions were asked during the interview in such a way as to allow the participant to express themselves in detail without any direction or comment. The interview was conducted individually by calling each woman by telephone. During the interview, the researcher transcribed the interviewee's sentences exactly as she expressed them. At the beginning of the analysis phase, the interview data were divided into sub-themes according to the main themes that had been determined beforehand in the researcher's notes. The working scheme of the qualitative research was applied in the seven stages of the interview technique defined by Kvale. The analysis technique was based on Gürbüz and Şahin's (2017) method of "data reduction, data labelling, creating categories and themes, revealing patterns, explaining and interpreting, and reporting", which was created by considering all the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being over
* 18 years of age,
* being mentally healthy,
* speaking Turkish,
* being in the earthquake zone during the earthquake. -

Exclusion Criteria:

* Refusing to participate in the study
* Having a language barrier to communication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Our study aims to examine the problems experienced by women after the earthquake
Study Population: The sample consisted of women aged 18 years and older who lived in Hatay, Kahramanmaraş and Adana provinces during and after the earthquake and who agreed to participate in the study.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | 10 minutes
  The first part of the form consists of personal information (age, occupation, marital status, number of children, spouse's occupation, educational status, income status).
  The second part consists of questions about changes experienced after the earthquake (loss of first-degree relatives, change in income status, living in a house/tent/container).
A semi-structured interview form | 30 minutes
  A semi-structured interview form, developed by the researcher through literature review, was used as a data collection tool. The third part consists of open-ended questions on opinions about life after the earthquake (changes in life in general; moving, changing jobs, etc.; problems of being a woman; hygiene, etc.).
  Study questions:
  * What are the demographic changes experienced by women after the earthquake?
  * What are the physical problems experienced by women after the earthquake?
  * What are the psychological/spiritual problems experienced by women after the earthquake?
  * What are the needs and difficulties of women after the earthquake?
  * What are the difficulties experienced by women in social life after the earthquake?
consists of questions about changes experienced after the earthquake | 10 minutes
  The second part consists of questions about changes experienced after the earthquake (loss of first-degree relatives, change in income status, living in a house/tent/container).
  The interview form consists of 18 questions, the last 5 of which are open questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ozeninam, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No